CLINICAL TRIAL: NCT01714219
Title: Effect of New Posterior Reconstruction Method on Recovery of Continence After Robot-assisted Laparoscopic Prostatectomy: Prospective, Single-blinded, Randomized Controlled Trial
Brief Title: Effect of New Posterior Reconstruction Method on Recovery of Continence After Robot-assisted Laparoscopic Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Sang Eun Lee, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNUBH-URO-2012-02
Record Dates: First submitted 2012-10-19; First posted 2012-10-25 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Localized Prostate Cancer; Urinary Incontinence
Keywords: prostatic neoplasms; prostatectomy; robotics; urinary incontinence
MeSH Terms: conditions — Urinary Incontinence; Prostatic Neoplasms | interventions — Posterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Posterior reconstruction (Experimental): * New posterior reconstruction, which entails opposition of the median dorsal fibrous raphe solely to the posterior counterpart of the detrusor apron
  * Vesicourethral anastomosis using the van Velthoven method
  * Anterior reconstruction, which involved opposing the anterior detrusor apron to the remaining puboprostatic ligaments and dorsal vascular complex
  Interventions: Procedure: Posterior reconstruction
- No posterior reconstruction (No Intervention): * No posterior reconstruction
  * Vesicourethral anastomosis using the van Velthoven method
  * Anterior reconstruction, which involved opposing the anterior detrusor apron to the remaining puboprostatic ligaments and dorsal vascular complex

INTERVENTIONS:
Procedure: Posterior reconstruction
  Arms: Posterior reconstruction

SUMMARY:
Incontinence is one of the most common complications of radical prostatectomy. The continence rate is not significantly improved even by robot-assisted laparoscopic prostatectomy (RALP). However, some reports suggested that posterior reconstruction (PR) behind vesicourethral anastomosis could improve early recovery of continence during open, laparoscopic or robot-assisted radical prostatectomy.

But, recent prospective studies reported no benefit of PR after RALP, which was the opposite result of those of previous studies. However the PR techniques used in these prospective studies seem to be quite different from the previous techniques. They seem to have used single-step PR, which opposes the median dorsal fibrous raphe (MDFR) only to the Denonvilliers' fascia (DF). By contrast, the original technique incorporated additional reconstruction between the MDFR and the posterior bladder wall 1-2 cm from the new bladder neck.

Our group identified this anatomic structure as the posterior counterpart of the detrusor apron (PDA). The PDA is a strong, thick functional tissue containing muscle that is more appropriate for pulling and fixing the MDFR than the DF. As such, we hypothesized that the key proximal structure for PR is not DF, but rather PDA. Furthermore, single-step reconstruction between MDFR and PDA could be enough for PR. We previously investigated whether our new PR technique, which entails opposition of the MDFR solely to the PDA, would improve continence recovery compared with the standard RALP technique without PR. And our retrospective study demonstrated that this new PR technique during RALP significantly shortens the time to the recovery of continence compared with the standard technique, which does not incorporate PR (Int J Urol, 2012;19:683-7).

Thus, we plan to validate this result by a well-designed, prospective, randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* pathologically proven localized prostate cancer (≤cT3a)
* patients to undergo robot-assisted laparoscopic prostatectomy by a single surgeon (Sang Eun Lee)

Exclusion Criteria:

* prior hormone therapy
* prior radiation treatment on prostate or pelvis
* preoperative urinary incontinence
* refused to participate

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Complete recovery of urinary continence | 6 months
  Duration of complete continence recovery defined as no pad use measured by question 5 of EPIC questionnaire.

SECONDARY OUTCOMES:
Duration of social continence recovery | 6 months
  Defined as 0 or 1 measured by EPIC question 5.
Continence score at 3 months | 3 months
  By EPIC question 5.
  * 0 vs. 1-3
  * mean value
Urinary leak at 3 months | 3 months
  By EPIC question 1,
  * 1-3 vs. 4-5
  * mean value
Self perception (QoL) of urinary function at 3 months | 3 months
  By EPIC question 7,
  * 0-1 vs. 2-4
  * mean value
Total operative time | At the day of surgery
  * Total operative time
  * Console time
Estimated blood loss | At the day of surgery
Complication | 6 months
  Complication by modified Clavien-Dindo grade

CONTACTS AND LOCATIONS:
Overall Officials: Sang Eun Lee, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea